CLINICAL TRIAL: NCT04942561
Title: Effect of Immersive Virtual Reality on Pain and Anxiety in Pediatric Peripheral Intravenous Catheter Access: A Randomized Clinical Trial
Brief Title: VR to Reduce Pain/Anxiety During IV Starts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: AppliedVR Inc. (Industry)
Responsible Party: Principal Investigator, Jeffrey I Gold, PhD, Principal Investigator, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHLA-15-00549_A
Record Dates: First submitted 2021-06-18; First posted 2021-06-28 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Radiology
Keywords: IV Stick; Pain; Anxiety; Virtual Reality; Radiology
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No VR) Randomization (No Intervention): In the standard of care treatment condition, participants will receive the standard CHLA treatment protocol for PIVC placement (i.e., a topical numbing spray and Buzzy® Bee, a vibrating device placed near the PIVC site for pain distraction).
- VR Randomization (Experimental): Children in the VR condition will undergo the invasive procedure while distracted by interaction with an immersive virtual environment (VE) presented via a head mounted display (HMD). The intervention group will receive standard CHLA treatment with VR distraction. Patients began gameplay <5 minutes before their PIVC placement and concluded after successful vascular access.
  Interventions: Device: Samsung Gear VR; Device: Merge VR

INTERVENTIONS:
Device: Samsung Gear VR — Participants 13 -21 years old can use the Samsung Gear VR. The VE is mobile based (Samsung with the Gear VR) and has active matrix LCDs with high pixel resolution, creating a bright, vibrant color and a quality image. Participants will engage with BearBlast (appliedVR™), a multi-sensory VR game in which users travel on a pre-set path through a colorful, highly-interactive 3-D environment filled with animated landscapes, buildings, and clouds, during which the user's gaze controls the direction of a firing cannon to knock down teddy bears. The VR game is equipped with a head-tracking system, enabling the player to look around the VE. Therefore, the child will be receiving distraction via 3-D visual and auditory sensory, thus supplying a multi-sensory immersive experience. While wearing these glasses, the children only can see the HMD screen so that the immersion and presence will be increased. The VR glasses will be sanitized before every use to minimize chance of infection.
  Arms: VR Randomization
Device: Merge VR — Participants 10-21 years can use the Merge. The VE to be used in this study is mobile based (Pixel with the Merge) and has active matrix LCDs with high pixel resolution, creating a bright, vibrant color and a quality image. Participants will engage with BearBlast (appliedVR™), a multi-sensory VR game in which users travel on a pre-set path through a colorful, highly-interactive 3-D environment filled with animated landscapes, buildings, and clouds, during which the user's gaze controls the direction of a firing cannon to knock down teddy bears. The VR game is equipped with a head-tracking system, enabling the player to look around the VE. Therefore, the child will be receiving distraction via 3-D visual and auditory sensory, thus supplying a multi-sensory immersive experience. While wearing these glasses, the children only can see the HMD screen so that the immersion and presence will be increased. The VR glasses will be sanitized before every use to minimize chance of infection.
  Arms: VR Randomization

SUMMARY:
This study aims to test the effectiveness of virtual reality (VR) as a non-pharmaceutical intervention to reduce pain and anxiety in children undergoing peripheral intravenous catheter (PIVC) access in the Department of Radiology and Imaging or the outpatient Infusion Center at CHLA, as measured by self- and proxy-report.

DETAILED DESCRIPTION:
Distraction is a form of non pharmacological intervention for reducing pain and anxiety in children during painful medical procedures (e.g., venipuncture, IV placement). Recent technological developments in the area of virtual reality (VR) provide new and potentially more effective ways of distracting children from the pain and anxiety associated with medical procedures. While initial studies of VR pain distraction are promising, few have studied the effectiveness of the technology in children, using a multi-method approach. The current study aims to recruit 115 children ages 10-21 years and their caregivers who arrive at the hospital for peripheral intravenous catheter (PIVC) access in the Department of Radiology and Imaging or the outpatient Infusion Center. Children and their parents will be randomly assigned to one of two treatment conditions: 1) existing hospital standard of care or 2) standard of care plus distraction via VR. Children and caregivers will be asked to complete measures assessing pain and anxiety both before and after the procedure. In addition, objective measures of child pain and distress during the PIVC access will be taken using coding of behavioral/verbal expressions. Univariate Analysis of Variance (ANOVA) will be used to compare differences in primary and secondary outcome variables in VR + standard of care to standard of care only conditions when pre and post-operative measures are available. Univariate ANOVA will be used to compare conditions on post-operative variables.

ELIGIBILITY:
Inclusion Criteria for Children:

1. Children who are 10-21 years old
2. Children who are English speaking (caregivers may be Spanish English speaking or Spanish speaking)
3. Children who are undergoing PIVC access in the Department of Radiology and Imaging or the outpatient Infusion Center.
4. Only children who are in the normal range of development will be recruited for this study. This will be assessed by report from the parents. The rationale for excluding patients with developmental delay is that due to their cognitive impairments, such children react to the stressors of surgery differently than do children without such developmental delay. It is unclear how such children would use the interventions included in this study, and it is likely that their responses on baseline and outcome measures will differ from children of normal developmental parameters.

Inclusion criteria for healthcare providers:

1. Healthcare providers must be 18 years old or older
2. Healthcare providers must be Children's Hospital Los Angeles staff
3. Healthcare providers may participate if they have witnessed and/or administered the medical procedure

Exclusion Criteria:

1. Children who are currently taking pain medication or anxiolytic medication will be excluded from this study.
2. Children with a psychiatric disorder, organic brain syndrome, mental retardation, or other known cognitive/neurological disorders
3. Children with visual, auditory, or tactile deficits that would interfere with the ability to complete the experimental tasks
4. Children with a history of seizure disorder.
5. Children currently sick with flu-like symptoms or experiencing a headache or earache.
6. Children with known or suspected motion sickness

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 107 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2019-07-24 (Actual); Study Completion 2019-07-24 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | Approximately 5 minutes to one hour before procedure
  The VAS anticipatory anxiety measure is a vertical VAS, anchored with 0 at the bottom indicating the least amount and 10 at the top indicating the greatest amount, in response to the instruction to rate "how nervous, afraid, or worried" they were about the upcoming task. The scale also has color cues, graded from yellow at the bottom to dark red at the top, as well as a neutral face at the bottom and a face showing a negative expression at the top. Prior research used the VAS to rate anticipatory anxiety and pain in children
Faces Pain Scale-Revised (FPS-R) | Approximately 5 minutes to one hour before procedure
  Revised is an updated version of the Wong-Baker Faces Pain Rating Scale depicting no pain as a neutral expression as compared with the smiling face of the original measure. The child is asked to point to the face cartoon that depicts how they are currently feeling because of their pain. Face measures are thought to measure pain intensity, and the Wong-Baker Faces measure has demonstrated good reliability and validity.

SECONDARY OUTCOMES:
Gold & Rizzo Immersion/Presence (GRIP) Inventory | Approximately 5 minutes to one hour before procedure
  Gold & Rizzo Immersion/Presence (GRIP) Inventory is a Child Presence Questionnaire was developed out of a content analysis of the entire domain of adult presence items and selection and adaptation of appropriate items for assessing the child's sense of believability of their experience. This 16-item measure is verbally administered to children and asks them to respond according to a 3-point Likert-like format. Items assess the child's sense of involvement, realism, and transportation into the experience. Patients in the VR condition will complete the Child Presence Questionnaire post-procedure to assess level of VR immersion.
Childhood Anxiety Sensitivity Index (CASI) | Approximately 5 minutes to one hour before procedure
  This 18-item measure utilizes a three-point Likert scale (none (1), some (2), a lot (3)) to assess how negatively patients view anxiety symptoms. Items are summed with a higher score indicating greater anxiety sensitivity.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey I Gold, PhD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gold JI, Mahrer NE. Is Virtual Reality Ready for Prime Time in the Medical Space? A Randomized Control Trial of Pediatric Virtual Reality for Acute Procedural Pain Management. J Pediatr Psychol. 2018 Apr 1;43(3):266-275. doi: 10.1093/jpepsy/jsx129. PMID 29053848
- [Background] Won AS, Bailey J, Bailenson J, Tataru C, Yoon IA, Golianu B. Immersive Virtual Reality for Pediatric Pain. Children (Basel). 2017 Jun 23;4(7):52. doi: 10.3390/children4070052. PMID 28644422
- [Background] Ahmadpour N, Keep M, Janssen A, Rouf AS, Marthick M. Design Strategies for Virtual Reality Interventions for Managing Pain and Anxiety in Children and Adolescents: Scoping Review. JMIR Serious Games. 2020 Jan 31;8(1):e14565. doi: 10.2196/14565. PMID 32012042
- [Background] Matsangidou M, Ang CS, Sakel M. Clinical utility of virtual reality in pain management: a comprehensive research review. Br J Neurosci Nurs. 2017;13(3):133-143. doi:10.12968/bjnn.2017.13.3.133
- [Background] Deacon B, Abramowitz J. Anxiety sensitivity and its dimensions across the anxiety disorders. J Anxiety Disord. 2006;20(7):837-57. doi: 10.1016/j.janxdis.2006.01.003. Epub 2006 Feb 8. PMID 16466904
- [Background] Kazak AE, Kassam-Adams N, Schneider S, Zelikovsky N, Alderfer MA, Rourke M. An integrative model of pediatric medical traumatic stress. J Pediatr Psychol. 2006 May;31(4):343-55. doi: 10.1093/jpepsy/jsj054. Epub 2005 Aug 10. PMID 16093522
- [Background] Inan G, Inal S. The Impact of 3 Different Distraction Techniques on the Pain and Anxiety Levels of Children During Venipuncture: A Clinical Trial. Clin J Pain. 2019 Feb;35(2):140-147. doi: 10.1097/AJP.0000000000000666. PMID 30362982
- [Background] Kucuk Alemdar D, Yaman Aktas Y. The Use of the Buzzy, Jet Lidokaine, Bubble-blowing and Aromatherapy for Reducing Pediatric Pain, Stress and Fear Associated with Phlebotomy. J Pediatr Nurs. 2019 Mar-Apr;45:e64-e72. doi: 10.1016/j.pedn.2019.01.010. Epub 2019 Jan 30. PMID 30711327
- [Background] Thrane SE, Wanless S, Cohen SM, Danford CA. The Assessment and Non-Pharmacologic Treatment of Procedural Pain From Infancy to School Age Through a Developmental Lens: A Synthesis of Evidence With Recommendations. J Pediatr Nurs. 2016 Jan-Feb;31(1):e23-32. doi: 10.1016/j.pedn.2015.09.002. Epub 2015 Sep 28. PMID 26424196
- [Background] Bandstra NF, Skinner L, Leblanc C, Chambers CT, Hollon EC, Brennan D, Beaver C. The role of child life in pediatric pain management: a survey of child life specialists. J Pain. 2008 Apr;9(4):320-9. doi: 10.1016/j.jpain.2007.11.004. Epub 2008 Jan 16. PMID 18201933
- [Background] Dumoulin S, Bouchard S, Ellis J, Lavoie KL, Vezina MP, Charbonneau P, Tardif J, Hajjar A. A Randomized Controlled Trial on the Use of Virtual Reality for Needle-Related Procedures in Children and Adolescents in the Emergency Department. Games Health J. 2019 Aug;8(4):285-293. doi: 10.1089/g4h.2018.0111. Epub 2019 May 24. PMID 31135178
- [Background] Uman LS, Chambers CT, McGrath PJ, Kisely S. A systematic review of randomized controlled trials examining psychological interventions for needle-related procedural pain and distress in children and adolescents: an abbreviated cochrane review. J Pediatr Psychol. 2008 Sep;33(8):842-54. doi: 10.1093/jpepsy/jsn031. Epub 2008 Apr 2. PMID 18387963
- [Background] Das DA, Grimmer KA, Sparnon AL, McRae SE, Thomas BH. The efficacy of playing a virtual reality game in modulating pain for children with acute burn injuries: a randomized controlled trial [ISRCTN87413556]. BMC Pediatr. 2005 Mar 3;5(1):1. doi: 10.1186/1471-2431-5-1. PMID 15745448
- [Background] Dunn A, Patterson J, Biega CF, Grishchenko A, Luna J, Stanek JR, Strouse R. A Novel Clinician-Orchestrated Virtual Reality Platform for Distraction During Pediatric Intravenous Procedures in Children With Hemophilia: Randomized Controlled Trial. JMIR Serious Games. 2019 Jan 9;7(1):e10902. doi: 10.2196/10902. PMID 30626567
- [Background] Furman E, Jasinevicius TR, Bissada NF, Victoroff KZ, Skillicorn R, Buchner M. Virtual reality distraction for pain control during periodontal scaling and root planing procedures. J Am Dent Assoc. 2009 Dec;140(12):1508-16. doi: 10.14219/jada.archive.2009.0102. PMID 19955069
- [Background] Gershon J, Zimand E, Pickering M, Rothbaum BO, Hodges L. A pilot and feasibility study of virtual reality as a distraction for children with cancer. J Am Acad Child Adolesc Psychiatry. 2004 Oct;43(10):1243-9. doi: 10.1097/01.chi.0000135621.23145.05. PMID 15381891
- [Background] Gold JI, Kim SH, Kant AJ, Joseph MH, Rizzo AS. Effectiveness of virtual reality for pediatric pain distraction during i.v. placement. Cyberpsychol Behav. 2006 Apr;9(2):207-12. doi: 10.1089/cpb.2006.9.207. PMID 16640481
- [Background] Hoffman HG, Patterson DR, Carrougher GJ, Sharar SR. Effectiveness of virtual reality-based pain control with multiple treatments. Clin J Pain. 2001 Sep;17(3):229-35. doi: 10.1097/00002508-200109000-00007. PMID 11587113
- [Background] Morris LD, Louw QA, Grimmer-Somers K. The effectiveness of virtual reality on reducing pain and anxiety in burn injury patients: a systematic review. Clin J Pain. 2009 Nov-Dec;25(9):815-26. doi: 10.1097/AJP.0b013e3181aaa909. PMID 19851164
- [Background] Schneider SM, Kisby CK, Flint EP. Effect of virtual reality on time perception in patients receiving chemotherapy. Support Care Cancer. 2011 Apr;19(4):555-64. doi: 10.1007/s00520-010-0852-7. Epub 2010 Mar 26. PMID 20336327
- [Background] Ashmore J, Di Pietro J, Williams K, Stokes E, Symons A, Smith M, Clegg L, McGrath C. A Free Virtual Reality Experience to Prepare Pediatric Patients for Magnetic Resonance Imaging: Cross-Sectional Questionnaire Study. JMIR Pediatr Parent. 2019 Apr 18;2(1):e11684. doi: 10.2196/11684. PMID 31518319
- [Background] Hua Y, Qiu R, Yao WY, Zhang Q, Chen XL. The Effect of Virtual Reality Distraction on Pain Relief During Dressing Changes in Children with Chronic Wounds on Lower Limbs. Pain Manag Nurs. 2015 Oct;16(5):685-91. doi: 10.1016/j.pmn.2015.03.001. Epub 2015 May 9. PMID 25972074
- [Background] Wiederhold BK, Gao K, Sulea C, Wiederhold MD. Virtual reality as a distraction technique in chronic pain patients. Cyberpsychol Behav Soc Netw. 2014 Jun;17(6):346-52. doi: 10.1089/cyber.2014.0207. PMID 24892196
- [Background] Neugebauer V, Li W, Bird GC, Han JS. The amygdala and persistent pain. Neuroscientist. 2004 Jun;10(3):221-34. doi: 10.1177/1073858403261077. PMID 15155061
- [Background] Chan E, Hovenden M, Ramage E, Ling N, Pham JH, Rahim A, Lam C, Liu L, Foster S, Sambell R, Jeyachanthiran K, Crock C, Stock A, Hopper SM, Cohen S, Davidson A, Plummer K, Mills E, Craig SS, Deng G, Leong P. Virtual Reality for Pediatric Needle Procedural Pain: Two Randomized Clinical Trials. J Pediatr. 2019 Jun;209:160-167.e4. doi: 10.1016/j.jpeds.2019.02.034. Epub 2019 Apr 29. PMID 31047650
- [Background] Walther-Larsen S, Petersen T, Friis SM, Aagaard G, Drivenes B, Opstrup P. Immersive Virtual Reality for Pediatric Procedural Pain: A Randomized Clinical Trial. Hosp Pediatr. 2019 Jul;9(7):501-507. doi: 10.1542/hpeds.2018-0249. Epub 2019 Jun 3. PMID 31160472
- [Background] Wong CL, Lui MMW, Choi KC. Effects of immersive virtual reality intervention on pain and anxiety among pediatric patients undergoing venipuncture: a study protocol for a randomized controlled trial. Trials. 2019 Jun 20;20(1):369. doi: 10.1186/s13063-019-3443-z. PMID 31221208
- [Background] Hicks CL, von Baeyer CL, Spafford PA, van Korlaar I, Goodenough B. The Faces Pain Scale-Revised: toward a common metric in pediatric pain measurement. Pain. 2001 Aug;93(2):173-183. doi: 10.1016/S0304-3959(01)00314-1. PMID 11427329
- [Background] Tomlinson D, von Baeyer CL, Stinson JN, Sung L. A systematic review of faces scales for the self-report of pain intensity in children. Pediatrics. 2010 Nov;126(5):e1168-98. doi: 10.1542/peds.2010-1609. Epub 2010 Oct 4. PMID 20921070
- [Background] Bringuier S, Dadure C, Raux O, Dubois A, Picot MC, Capdevila X. The perioperative validity of the visual analog anxiety scale in children: a discriminant and useful instrument in routine clinical practice to optimize postoperative pain management. Anesth Analg. 2009 Sep;109(3):737-44. doi: 10.1213/ane.0b013e3181af00e4. PMID 19690240
- [Background] Silverman WK, Fleisig W, Rabian B, Peterson RA. Child Anxiety Sensitivity Index. J Clin Child Psychol. 1991;20(2):162-168. doi:10.1207/s15374424jccp2002_7
- [Background] Felitti VJ, Anda RF, Nordenberg D, Williamson DF, Spitz AM, Edwards V, Koss MP, Marks JS. Relationship of childhood abuse and household dysfunction to many of the leading causes of death in adults. The Adverse Childhood Experiences (ACE) Study. Am J Prev Med. 1998 May;14(4):245-58. doi: 10.1016/s0749-3797(98)00017-8. PMID 9635069
- [Background] Spiegel B, Fuller G, Lopez M, Dupuy T, Noah B, Howard A, Albert M, Tashjian V, Lam R, Ahn J, Dailey F, Rosen BT, Vrahas M, Little M, Garlich J, Dzubur E, IsHak W, Danovitch I. Virtual reality for management of pain in hospitalized patients: A randomized comparative effectiveness trial. PLoS One. 2019 Aug 14;14(8):e0219115. doi: 10.1371/journal.pone.0219115. eCollection 2019. PMID 31412029
- [Background] Tashjian VC, Mosadeghi S, Howard AR, Lopez M, Dupuy T, Reid M, Martinez B, Ahmed S, Dailey F, Robbins K, Rosen B, Fuller G, Danovitch I, IsHak W, Spiegel B. Virtual Reality for Management of Pain in Hospitalized Patients: Results of a Controlled Trial. JMIR Ment Health. 2017 Mar 29;4(1):e9. doi: 10.2196/mental.7387. PMID 28356241
- [Background] Vadivelu N, Kai AM, Kodumudi V, Sramcik J, Kaye AD. The Opioid Crisis: a Comprehensive Overview. Curr Pain Headache Rep. 2018 Feb 23;22(3):16. doi: 10.1007/s11916-018-0670-z. PMID 29476358
- [Background] Amin AM, Tong X, Gromala D, Shaw CD. Cardboard Mobile Virtual Reality as an Approach for Pain Distraction in Clinical Settings: Comparison, Exploration and Evaluation with Oculus Rift. In: Proceedings of the 2017 CHI Conference Extended Abstracts on Human Factors in Computing Systems. CHI EA '17. Association for Computing Machinery; 2017:2345-2351. doi:10.1145/3027063.3053234
- [Background] Hendricks TM, Gutierrez CN, Stulak JM, Dearani JA, Miller JD. The Use of Virtual Reality to Reduce Preoperative Anxiety in First-Time Sternotomy Patients: A Randomized Controlled Pilot Trial. Mayo Clin Proc. 2020 Jun;95(6):1148-1157. doi: 10.1016/j.mayocp.2020.02.032. PMID 32498771
- [Background] Ahmadpour N, Randall H, Choksi H, Gao A, Vaughan C, Poronnik P. Virtual Reality interventions for acute and chronic pain management. Int J Biochem Cell Biol. 2019 Sep;114:105568. doi: 10.1016/j.biocel.2019.105568. Epub 2019 Jul 12. PMID 31306747
- [Background] Gershon J, Zimand E, Lemos R, Rothbaum BO, Hodges L. Use of virtual reality as a distractor for painful procedures in a patient with pediatric cancer: a case study. Cyberpsychol Behav. 2003 Dec;6(6):657-61. doi: 10.1089/109493103322725450. PMID 14756933
- [Background] Firoozabadi R, Elhaddad M, Drever S, Soltani M, Githens M, Kleweno CP, Sharar SR, Patterson DR, Hoffman HG. Case Report: Virtual Reality Analgesia in an Opioid Sparing Orthopedic Outpatient Clinic Setting: A Case Study. Front Virtual Real. 2020 Dec;1:553492. doi: 10.3389/frvir.2020.553492. Epub 2020 Dec 14. PMID 33585832
- [Background] Ozalp Gerceker G, Ayar D, Ozdemir EZ, Bektas M. Effects of virtual reality on pain, fear and anxiety during blood draw in children aged 5-12 years old: A randomised controlled study. J Clin Nurs. 2020 Apr;29(7-8):1151-1161. doi: 10.1111/jocn.15173. Epub 2020 Jan 22. PMID 31889358
- [Background] Thomas JJ, Albietz J, Polaner D. Virtual reality for lumbar puncture in a morbidly obese patient with leukemia. Paediatr Anaesth. 2018 Nov;28(11):1059-1060. doi: 10.1111/pan.13505. Epub 2018 Oct 4. PMID 30284748
- [Background] Wong CL, Li CK, Chan CWH, Choi KC, Chen J, Yeung MT, Chan ON. Virtual Reality Intervention Targeting Pain and Anxiety Among Pediatric Cancer Patients Undergoing Peripheral Intravenous Cannulation: A Randomized Controlled Trial. Cancer Nurs. 2021 Nov-Dec 01;44(6):435-442. doi: 10.1097/NCC.0000000000000844. PMID 32511154
- [Background] Loreto-Quijada D, Gutierrez-Maldonado J, Gutierrez-Martinez O, Nieto R. Testing a virtual reality intervention for pain control. Eur J Pain. 2013 Oct;17(9):1403-10. doi: 10.1002/j.1532-2149.2013.00316.x. Epub 2013 Apr 12. PMID 23580493
- [Background] Piskorz J, Czub M. Effectiveness of a virtual reality intervention to minimize pediatric stress and pain intensity during venipuncture. J Spec Pediatr Nurs. 2018 Jan;23(1). doi: 10.1111/jspn.12201. Epub 2017 Nov 20. PMID 29155488